CLINICAL TRIAL: NCT00888251
Title: A Multicenter, Retrospective Study to Evaluate the Effectiveness of the OPTIFAST Weight Management Program
Brief Title: Evaluation of a Weight Management Program
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 08.27.CLI
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Obesity
Keywords: Obesity; Meal replacement; Obesity treatment; Weight management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Comprehensive weight management program
  Interventions: Other: Comprehensive weight management program

INTERVENTIONS:
Other: Comprehensive weight management program — Full meal replacement, behaviorial modification, medical monitoring, exercise.
  Other Names: OPTIFAST Program

SUMMARY:
This retrospective chart review and data abstraction will evaluate and quantify the effectiveness of a comprehensive weight management program. The hypothesis is that the program will positively affect weight, weight-related comorbidities and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Records of the first 40 study center participants who enrolled in the OPTIFAST Program from January 1, 2006 through June 30, 2006
* Records of subjects who completed the active weight loss phase of the program
* Records where data is available through the transitional phase of the program

Exclusion Criteria:

* Concurrent use of appetite suppressants or other weight loss medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OPTIFAST Program participants
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lutheran Weight Management Center, Fort Wayne, Indiana
  - Mercy Center for Weight Reduction, Des Moines, Iowa
  - Sparrow Weight Management Center, East Lansing, Michigan
  - Jewish Hospital Weight Management Center, Cincinnati, Ohio